CLINICAL TRIAL: NCT02601261
Title: How Anxiety in Pregnant Hospitalized Women Change wIth Internet Use
Acronym: HAWAII
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Collaborators: Azienda Ospedaliero Universitaria, Santa Maria della Misericordia di Udine, Italy (Other); Azienda Per I Servizi Sanitari N. 6 Friuli Occidentale (Other)
Responsible Party: Principal Investigator, Dario Gregori, Professor, University of Padova
Other Study IDs: HAWAII
Record Dates: First submitted 2015-10-29; First posted 2015-11-10 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Pregnant Women in All Gestational Ages Hospitalized for a Problem of Pregnancy
Keywords: pregnant; gestational ages; hospitalized; problem of pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with some access to internet during stay
  Interventions: Other: At the first day of hospitalization the field investigator will submit to pregnant women in a pathological condition five questionnaires
- Patients without access to internet during stay
  Interventions: Other: At the first day of hospitalization the field investigator will submit to pregnant women in a pathological condition five questionnaires

INTERVENTIONS:
Other: At the first day of hospitalization the field investigator will submit to pregnant women in a pathological condition five questionnaires — Some of these questionnaires will have to be completed every day and others every other day:
  1. The Internet questionnaire is divided in two parts. The first one investigates the use of internet at home and it will be administered only once, the second part will investigate the internet use at the hospital, in the case the women have a personal smartphone, tablet or personal computer (they are the owners) and it will be administered every other days.
  2. The questionnaire is aimed to understand the quality of life (EQ-5D) will be administered only once, at the beginning of the hospitalization.
  3. The STAI questionnaire is divided in to parts, the first part aims to determinate the state anxiety and it will be administered every other day, while the second part will discuss the anxiety itself, and has to completed only once.
  4. The short questionnaire on critical events occurring during the day,
  5. The short questionnaire with obstetric anamnesis.

SUMMARY:
Investigating the influence of Internet use to the level of state anxiety in hospitalized women with pathological pregnancy.

A recent research shown that the prevalence of antenatal anxiety changes during pregnancy at first trimester is 36.3%; the rate dropped to 32.3% at second trimester but increased again to 35.8% at third trimester (art. 29).According to the World Health Organization, mental health disorders are the leading cause of disease burden in woman from 15 to 44 years (art.6). A Swedish study indicated that the incidence of moderate or extreme symptoms of anxiety and depression of pregnant woman during the first trimester is 15,6% (art. 3).

DETAILED DESCRIPTION:
WHAT CAUSES ANXIETY IN PREGNANT WOMEN

Anxiety during pregnancy may expose the woman to a higher risk of a negative outcome in four different fields:

1. Fetal obstetric outcomes; 2. Neonatal outcomes; 3. Child development; 4. Risk to the woman.

1. The anxiety in pregnant woman may expose the fetus to a higher risk of spontaneous early labor, preterm delivery, lower birth weight, fetal distress, fetal growth restriction, risk for spontaneous abortion, risk of pre-eclampsia and for operative/instrumental deliveries. Furthermore could be a major risk for the uterine artery to have high resistance that could reduce blood flow to the fetus.
2. The neonates that had a mother with anxiety issues during pregnancy may have an higher risk of admission to neonatal ICU, have a lower Apgar score and small head circumference, growth retardation, slowed mental development and excessive crying, irritability, hostility and erratic sleep. The mother anxiety could also increase the possibility to have colic in the neonatal age.
3. On the other hand the maternity anxiety could have long-term negative effects on the child development. There are risks of negative effect on maternal-infant bonding, difficult with affect regulations, cognitive delays, behavioral and emotional difficulties, maladaptive and social interactions, cognitive delays, behavioral and emotional difficulties and maladaptive social interactions. Furthermore, the child could develop a major level of fear and anxiety during life, an insecure and disorganized attachment and lower IQ at age 15-15 years. Anxiety of the mothers during pregnancy could cause a non-optimal neuromotorial development of the child, a research demonstrated an association between the anxiety of the mother in late pregnancy and the infant behavior, his emotional problems and his difficult temperament during later infancy. To demonstrated the correlation between anxiety and negative outcomes during childhood a Belgian/Dutch study showed that the 14-15 years old person that had a mother with anxiety disorders reveals a major risk of impulsivity and cognitive disorders. Another study demonstrated the connection between antenatal anxiety and behavioral/emotional problems of a four years old child. Another probable negative outcome of the pregnant anxiety is the asthma during childhood. A study demonstrated that the baby with a anxious mother has an higher risk to the use of antibiotic, to have respiratory and skin illnesses in the first year of the life than the child born from a mother without anxiety disorder.
4. It is very important underline to that anxiety during pregnancy has a negative effect not only on the fetus and child but also on the mother as well. Many researches demonstrated a link between prenatal anxiety and postpartum depression, psychiatric complications, and a higher risk of preeclampsia. In addition, the mother suffering of anxiety requires more examination from an obstetrician and most of all require an elective caesarean section. Other negative outcomes are poor nutrition, impaired self-care of the mother, failure to follow medical and prenatal guidelines, and major exposure to use alcohol, drugs and tobacco.

INTERNET INFORMATION In 2004 the 4,5% of the researches of internet were about medical information and, in 2009, the 61% of adult Internet users in the United States searched for health-related information. The Internet allows people to have an immediately health information and also pregnant woman search information about pregnancy and connected problems. For example women affected with nausea and vomiting during early pregnancy search online how this problem could be treated. On the other hand, not all information available on the Internet are regulated, nor are always reliable or current.

ELIGIBILITY:
Inclusion Criteria:

* Italian speaking and reading ability;
* Age > 18 years
* Been hospitalized for a pathological pregnancy condition;
* Having a twin pregnancy;
* All gestational ages;
* Having been transferred from other hospitals.

Exclusion Criteria:

* Been under stressful family events (deaths, recent separation: self-reported)
* With a diagnosis of a mental psychiatric diseases;
* With a diagnosis of cancer pathology.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study has been powered to detect a difference on the average STAI state score (range 20-80) of 6 points between women with some access to internet during stay (at least 10 minutes/days of web browsing, besides e-mails) and those no accessing internet during stay. Assuming a Standard Deviation of the difference in STAI scores of about 8 points (art. 30-art. 33), and assuming that the ratio between the rate of women not using internet and that of women using internet is 0,42 (art. 31-art. 32) for specified alpha = 0.025 and power (1 - beta) of 90.0% a total of 109 women must be recruited (using a two-sample t-test with unknown variance).
  Data entry will be based on e-CRF running on the REDCAP Clinical Data Management System of the Service for Clinical Trials and Biometrics (Department of Cardiology, Thoracic and Vascular Sciences, University of Padova).
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
The association between the use of Internet and the level of anxiety in pregnant hospitalized women. | 10 days
  During the first day of hospitalization, the field investigator administers to every patient participating to the study all five questionnaires and on each questionnaire, it will be indicated the day when it has been completed.
  The study measures the level of state anxiety in hospitalized women with pathological pregnancy, influenced by internet use. The STAI questionnaire that evaluate the level of anxiety, is divided in to parts: the first part aims to determinate the state anxiety and it will be administered every other day, while the second part will discuss the anxiety itself, and has to completed only once.

SECONDARY OUTCOMES:
Using STAI questionnaire to evaluate how the level of anxiety changes during the hospitalization, in women with pathological pregnancy. | 10 days
Using Internet questionnaire to determinate the type of health information pregnant women are seeking online during and before the hospitalization and the number of them | 10 days
STAI questionnaire and Internet questionnaire used to compare the anxiety levels and the access to online health information between different subcategories: women having internet access during hospitalization and those who have not. | 10 days

REFERENCES:
- [Background] Rubertsson C, Hellstrom J, Cross M, Sydsjo G. Anxiety in early pregnancy: prevalence and contributing factors. Arch Womens Ment Health. 2014 Jun;17(3):221-8. doi: 10.1007/s00737-013-0409-0. Epub 2014 Jan 18. PMID 24442712
- [Background] van Batenburg-Eddes T, de Groot L, Huizink AC, Steegers EA, Hofman A, Jaddoe VW, Verhulst FC, Tiemeier H. Maternal symptoms of anxiety during pregnancy affect infant neuromotor development: the generation R study. Dev Neuropsychol. 2009;34(4):476-93. doi: 10.1080/87565640902964508. PMID 20183712
- [Background] Field T, Diego M, Hernandez-Reif M, Figueiredo B, Deeds O, Ascencio A, Schanberg S, Kuhn C. Comorbid depression and anxiety effects on pregnancy and neonatal outcome. Infant Behav Dev. 2010 Feb;33(1):23-9. doi: 10.1016/j.infbeh.2009.10.004. Epub 2009 Nov 27. PMID 19945170
- [Background] Fishell A. Depression and anxiety in pregnancy. J Popul Ther Clin Pharmacol. 2010 Fall;17(3):e363-9. Epub 2010 Oct 26. PMID 21041870
- [Background] O'Connor TG, Heron J, Golding J, Beveridge M, Glover V. Maternal antenatal anxiety and children's behavioural/emotional problems at 4 years. Report from the Avon Longitudinal Study of Parents and Children. Br J Psychiatry. 2002 Jun;180:502-8. doi: 10.1192/bjp.180.6.502. PMID 12042228
- [Background] Austin MP, Hadzi-Pavlovic D, Leader L, Saint K, Parker G. Maternal trait anxiety, depression and life event stress in pregnancy: relationships with infant temperament. Early Hum Dev. 2005 Feb;81(2):183-90. doi: 10.1016/j.earlhumdev.2004.07.001. PMID 15748973
- [Background] Van den Bergh BR, Marcoen A. High antenatal maternal anxiety is related to ADHD symptoms, externalizing problems, and anxiety in 8- and 9-year-olds. Child Dev. 2004 Jul-Aug;75(4):1085-97. doi: 10.1111/j.1467-8624.2004.00727.x. PMID 15260866
- [Background] O'Connor TG. Annotation: The 'effects' of parenting reconsidered: findings, challenges, and applications. J Child Psychol Psychiatry. 2002 Jul;43(5):555-72. doi: 10.1111/1469-7610.00046. PMID 12120853
- [Background] Beijers R, Jansen J, Riksen-Walraven M, de Weerth C. Maternal prenatal anxiety and stress predict infant illnesses and health complaints. Pediatrics. 2010 Aug;126(2):e401-9. doi: 10.1542/peds.2009-3226. Epub 2010 Jul 19. PMID 20643724
- [Background] Gao LL, Larsson M, Luo SY. Internet use by Chinese women seeking pregnancy-related information. Midwifery. 2013 Jul;29(7):730-5. doi: 10.1016/j.midw.2012.07.003. Epub 2012 Sep 5. PMID 22958935
- [Background] Lee AM, Lam SK, Sze Mun Lau SM, Chong CS, Chui HW, Fong DY. Prevalence, course, and risk factors for antenatal anxiety and depression. Obstet Gynecol. 2007 Nov;110(5):1102-12. doi: 10.1097/01.AOG.0000287065.59491.70. PMID 17978126
- [Background] Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S467-72. doi: 10.1002/acr.20561. No abstract available. PMID 22588767
- [Background] Minto C, Bauce B, Calore C, Rigato I, Folino F, Soriani N, Hochdorn A, Iliceto S, Gregori D. Is Internet use associated with anxiety in patients with and at risk for cardiomyopathy? Am Heart J. 2015 Jul;170(1):87-95, 95.e1-4. doi: 10.1016/j.ahj.2015.02.024. Epub 2015 Apr 9. PMID 26093868
- [Result] Ibanez G, Charles MA, Forhan A, Magnin G, Thiebaugeorges O, Kaminski M, Saurel-Cubizolles MJ; EDEN Mother-Child Cohort Study Group. Depression and anxiety in women during pregnancy and neonatal outcome: data from the EDEN mother-child cohort. Early Hum Dev. 2012 Aug;88(8):643-9. doi: 10.1016/j.earlhumdev.2012.01.014. Epub 2012 Feb 22. PMID 22361259